CLINICAL TRIAL: NCT04809012
Title: An Open-label, Multicenter, Phase 2 Basket Study to Investigate the Efficacy, Safety, Pharmacokinetics and Pharmacodynamics of STI-3031 in Patients With Selected Relapsed or Refractory Solid Tumors
Brief Title: Study of STI-3031 in Patients With Selected Relapsed or Refractory Solid Tumors
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Intended to be replaced with another Protocol
Sponsor: Sorrento Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PDL1-RRST-201
Record Dates: First submitted 2021-03-13; First posted 2021-03-22 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Solid Tumor; Refractory Tumor; Relapsed Solid Tumor
Keywords: PDL-1; RRST
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- STI-3031 (Experimental): 20 mg/kg STI-3031 administered intravenously Q2W
  Interventions: Biological: STI-3031

INTERVENTIONS:
Biological: STI-3031 — STI-3031 is an anti-PD-L1 antibody

SUMMARY:
This study evaluates the efficacy of STI-3031, an anti-PD-L1 antibody, in previously treated patients with selected solid tumors.

DETAILED DESCRIPTION:
This is an open-label, multicenter, Phase 2 basket study to investigate the efficacy, safety, pharmacokinetics and pharmacodynamics of STI-3031, an anti-PD-L1 antibody, in patients with selected RRSTs. All participants will receive STI-3031 20 mg/kg every 2 weeks (Q2W) via IV infusion over approximately 60 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score ≤ 2
* Has histologically- or cytologically-confirmed relapsing or refractory solid tumor and subject has exhausted all approved options that may, in the investigator's opinion, produce clinical benefit.
* Has at least one measurable disease per RECIST 1.1
* May have been treated with radiation therapy (RT) provided there is measurable disease outside the field of RT. Prior systemic RT must be completed at least 4 weeks before the first dose of study intervention. Prior focal radiotherapy must be completed at least 2 weeks before the first dose of study intervention. No radiopharmaceuticals are permitted within 8 weeks before the first dose of study intervention.
* Life expectancy of at least 16 weeks per investigator assessment
* Must have adequate hematologic, hepatic and renal function as assessed by specific laboratory criteria
* Willing to sign the informed consent form and comply with the study schedule and all other protocol requirements
* Females of childbearing potential (FCBP) must have a negative pregnancy test during the Screening Period prior to treatment. All heterosexually active FCBP and all heterosexually active male patients must agree to use effective double barrier methods of birth control throughout the study.
* At time of the first dose of study intervention, at least 14 days or 5 half-lives, whichever is shorter, since the last chemotherapy, immunotherapy, biological or investigational therapy, and have recovered from toxicities associated with such treatment to < Grade 2.

Exclusion Criteria:

* Previously treated with an anti-PD-L1 or anti-PD-1 antibody
* Known presence of symptomatic central nervous system (CNS) metastases unless considered adequately treated and off corticosteroids and/or anticonvulsant therapy for at least 2 weeks prior to first dose of study intervention.
* Prior allogeneic hematopoietic stem cell transplantation (HSCT) or solid organ transplantation. Prior autologous HSCT is allowed.
* Any other malignancy, excluding basal or squamous cell carcinoma of the skin, cervical carcinoma in situ, or localized prostate cancer, from which the participant has not been disease-free for at least 2 years.
* Any active autoimmune disease requiring treatment within the past 3 months or a documented history of autoimmune disease, or history of syndrome that required systemic steroids or immunosuppressive medications, except for participants with vitiligo, hormone replacement therapy for stable thyroid diseases and Type 1 diabetes mellitus.
* Evidence of active or latent tuberculosis (TB) infection
* Known viral infection with COVID-19, hepatitis B virus (HBV) hepatitis C virus (HCV), unless participant, as applicable, is negative on RT-PCR or rapid antigen tests, has been vaccinated, and has completed curative antiviral treatment and viral load is below the limit of quantification.
* Known active viral infection with human immunodeficiency virus (HIV)
* Active infection (viral, bacterial, or fungal) requiring intravenous (IV) systemic therapy within 14 days prior to the first dose of study intervention.
* Evidence of bleeding diathesis or coagulopathy.
* Conditions requiring chronic steroid use (> 10 mg/day of prednisone or equivalent).
* Recent history of attenuated viral vaccination within 30 days prior to the first dose of study intervention.
* Herbal preparations/medications are not allowed throughout the treatment period unless first discussed with and approved by the Medical Monitor.
* History of severe hypersensitivity reactions to other monoclonal antibodies or known hypersensitivity to the study intervention or its excipients.
* Known current drug or alcohol abuse
* Major surgical procedures ≤ 28 days prior to the first dose of study intervention, or minor surgical procedures ≤ 7 days prior to the first dose of study intervention. No waiting is required following port-a-catch placement or similar venous access device.
* Pregnant or lactating or intending on either during the study
* Severe or uncontrolled cardiac disease requiring treatment, congestive heart failure NYHA III or IV, unstable angina pectoris even if medically controlled, history of myocardial infarction during the last 3 months, serious arrhythmias requiring medication (with exception of atrial fibrillation or paroxysmal supraventricular tachycardia).
* Underlying medical conditions that, in the Investigator's opinion, will make the administration of study intervention hazardous or obscure the interpretation of toxicity determination or AEs, including psychiatric illness or social situation that would preclude study compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Baseline through study completion at up to approximately 3 years
  Objective response rate (ORR) as assessed using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria

SECONDARY OUTCOMES:
Safety as assessed by incidence and severity of adverse events | Baseline through study completion at up to approximately 3 years
  Incidence of treatment-emergent adverse events and their relationships to STI-3031
Duration of Response | Baseline through study completion at up to approximately 3 years
  Duration of response (DOR) as assessed using RECIST 1.1
Complete response rate and duration | Baseline through study completion at up to approximately 3 years
  Complete response (CR) rate and duration of CR as assessed using RECIST 1.1
Progression-Free Survival | Baseline through study completion at up to approximately 3 years
  Progression-free survival (PFS) and 12-month PFS as assessed using RECIST 1.1
Event-free survival | Baseline through study completion at up to approximately 3 years
  Event-free survival (EFS) as assessed using RECIST 1.1
Overall survival | Baseline through study completion at up to approximately 3 years
  Overall survival (OS) as assessed using RECIST 1.1
Time to next treatment | Baseline through study completion at up to approximately 3 years
  Time to next treatment (TTNT)
Incidence of anti-drug antibody | Baseline through study completion at up to approximately 3 years
  Incidence of anti-drug antibody (ADA) and correlation with exposure and activity as measured using serum titers of anti-STI-3031 antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Mike Royal, MD, Study Director — Sorrento Therapeutics